CLINICAL TRIAL: NCT00083187
Title: A Phase II Study of VNP40101M For Patients With Acute Myelogenous Leukemia Or High-Risk Myelodysplasia
Brief Title: VNP40101M in Treating Patients With Acute Myelogenous Leukemia or High-Risk Myelodysplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vion Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: VION-CLI-033; CDR0000365510 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2008-08

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative; chronic myelomonocytic leukemia; myelodysplastic/myeloproliferative neoplasm, unclassifiable; secondary myelodysplastic syndromes; de novo myelodysplastic syndromes; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Congenital Abnormalities | interventions — Hydroxyurea; laromustine

INTERVENTIONS:
Drug: hydroxyurea
Drug: laromustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as VNP40101M and hydroxyurea, work in different ways to stop cancer cells from dividing so they stop growing or die. Hydroxyurea may help VNP40101M kill more cancer cells by making cancer cells more sensitive to the drug.

PURPOSE: This phase II trial is studying how well giving VNP40101M with hydroxyurea works in treating patients with acute myelogenous leukemia or high-risk myelodysplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete response rate to VNP40101M in patients with acute myelogenous leukemia or high-risk myelodysplasia .
* Determine the toxic effects of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is an open-label, multicenter study. Patients are stratified to acute myelogenous leukemia (AML) or high risk myelodysplasia (MDS) patients ≥ 60 years old with no prior treatment vs AML patients any age in first relapse. (AML patients any age in first relapse closed to accrual 06/09/05).

Patients receive VNP40101M IV over 30 minutes once on day 1 (course 1).

Four to five weeks after the first course, patients undergo bone marrow aspiration and biopsy. If the bone marrow is improved but contains residual leukemia, patients receive a second course of VNP40101M (at the same dose as in course 1). If patients achieve complete response (CR), or partial CR after the first or second course, a consolidation course may be given comprising VNP40101M at a reduced dose.

Patients are followed monthly for 6 months, every 2 months for 12 months, and then every 3 months for 18 months .

PROJECTED ACCRUAL: A total of 230 patients (100 with acute myelogenous leukemia (AML) or high-risk myelodysplasia and 130 with AML in first relapse) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Acute myelogenous leukemia (AML), meeting the following criteria:

    * In first relapse after first treatment-induced complete remission (CR) (closed to accrual as of 06/09/05)

      * Duration of first CR less than 12 months
      * No prior treatment for first relapse except hydroxyurea
    * FAB type M0, M1, M2, M4-7
    * No acute promyelocytic leukemia
    * No prior treatment with a standard induction regimen containing cytotoxic agents* (for patients 60 years of age or older)
  * High-risk myelodysplasia, meeting the following criteria:

    * 60 years of age and over
    * No prior cytotoxic chemotherapy* except hydroxyurea
    * Prior gemtuzumab ozogamicin allowed
    * High risk defined as International Prognostic Scoring System score ≥ 1.5, defined by cytogenetics, % marrow blasts, and lineage cytopenias NOTE: *Prior low-dose, single-agent cytarabine, decitabine, or azacitidine not considered prior cytotoxic chemotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* ALT or AST ≤ 5 times upper limit of normal
* Chronic hepatitis allowed

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* No myocardial infarction within the past 3 months
* No symptomatic coronary artery disease
* No uncontrolled arrhythmias
* No uncontrolled congestive heart failure
* No other active heart disease

Other

* No uncontrolled active infection
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Up to 4 leukapheresis procedures allowed during the first 15 days of study treatment

Chemotherapy

* See Disease Characteristics
* Concurrent additional hydroxyurea (maximum dose of 5 g daily for up to 4 days) allowed between days 4 and 15 of each study course to control elevated blast levels

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Recovered from all prior therapy
* At least 72 hours since prior anti-leukemic treatment with a non-cytotoxic agent
* No concurrent disulfiram (Antabuse)
* No other concurrent anticancer drugs except anagrelide within the first 15 days of study treatment to control elevated platelet counts
* No other concurrent treatment for leukemia, except hydroxyurea used during study treatment
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2005-11; Primary Completion 2007-01 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Complete response rate
Toxic effects
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Francis J. Giles, MD, Study Chair — M.D. Anderson Cancer Center
Locations (5):
- United States (3):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
- Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille, France
- King's College Hospital, London, England, United Kingdom

REFERENCES:
- [Result] Gerson SL, Karp J, Rizzieri D, et al.: Low levels of pre-treatment O6-alkylguanine transferase (AGT) in patients with AML correlate with response to Cloretazine® (VNP40101M) induction therapy. [Abstract] American Association for Cancer Research: 98th Annual Meeting, April 14-18, 2007, Los Angeles, CA. A-2640, 2007.
- [Result] Giles F, Rizzieri D, Karp J, Vey N, Ravandi F, Faderl S, Khan KD, Verhoef G, Wijermans P, Advani A, Roboz G, Kantarjian H, Bilgrami SF, Ferrant A, Daenen SM, Karsten V, Cahill A, Albitar M, Mufti G, O'Brien S. Cloretazine (VNP40101M), a novel sulfonylhydrazine alkylating agent, in patients age 60 years or older with previously untreated acute myeloid leukemia. J Clin Oncol. 2007 Jan 1;25(1):25-31. doi: 10.1200/JCO.2006.07.0961. Epub 2006 Dec 4. PMID 17146105